CLINICAL TRIAL: NCT03106480
Title: Diabetes and Associated Complications in HIV Patients
Brief Title: Diabetes Mellitus and HIV Study in Mwanza
Acronym: CICADA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other); London School of Hygiene and Tropical Medicine (Other); University of Bergen (Other); Vanderbilt University (Other); Tanzania Commission for AIDS, Tanzania (Unknown); Hindu Mandal Hospital,Tanzania (Unknown)
Responsible Party: Principal Investigator, Dr George PrayGod, Principal Research Scientist, National Institute for Medical Research, Tanzania
Other Study IDs: 16-P01-TAN
Record Dates: First submitted 2017-02-15; First posted 2017-04-10 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus; HIV/AIDS
Keywords: Pre-diabetes; Diabetes Mellitus; HIV; ART; Body composition; Inflammation; Insulin resistance; Beta-cell function; Pre-Hypertension; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Acquired Immunodeficiency Syndrome; Glucose Intolerance; Inflammation; Insulin Resistance; Prehypertension; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV and Diabetes Cohort: Participants recruited in the study will have diverse characteristics. Participants will either be HIV infected or HIV negative and among those HIV-infected there will be those on ART and those not on ART. In addition, participants will have other background characteristics like having history of tuberculosis treatment, being malnourished while starting ART, having diabetes at ART initiation etc. Investigators will also be able to examine the effect of immune activation, body composition changes, and other related factors on the risk of diabetes. This diversity of characteristics will help provide adequate data to address study outcomes.

SUMMARY:
Emerging evidence from high-income countries suggests that diabetes mellitus is become a major health problem among HIV-infected patients. However, due to differences in social, environmental, and genetic factors data from high-income countries can not be extrapolated directly to low-income countries. This study investigates HIV, ART, inflammation, and body composition changes as risk factors for diabetes mellitus among HIV-infected patients in Tanzania.

DETAILED DESCRIPTION:
Access to antiretroviral therapy (ART) is increasing rapidly in low-income countries and HIV-infected patients initiate ART much earlier. As a result, these patients have prolonged life spans and, hence, longer HIV and ART exposure. Emerging data from developed countries suggest that HIV-infected patients have a higher risk than HIV-uninfected people of developing diabetes mellitus (DM) and other non-communicable diseases. The excess diabetes risk is probably related to multiple factors including HIV-associated inflammation, the use of some antiretroviral therapy (ART) regimens, and body composition changes associated with HIV and ART. As a result, HIV-infected populations may develop DM at a younger age and may have a higher mortality if management is not optimal as may be the case in resource-limited countries of Sub-Saharan Africa (SSA).

Most of the data to-date on HIV and DM are from high-income countries, and data in SSA are few and inconsistent. Because of differences in genetic composition as well as environmental factors including high burden of infectious diseases in resource-limited settings, data from high-income countries cannot be extrapolated and reliably used to improve quality of DM care among HIV patients in SSA. The objective of this study is to investigate if HIV, ART, and body composition changes occurring during ART use are associated with higher risk of DM as well as other risk factors for cardiovascular diseases in Tanzanian patients, and examine if HIV increases the risk of DM associated complications. This study is funded by the Danish Ministry of Foreign Affairs from 2016 to 2021.

ELIGIBILITY:
Inclusion Criteria:

* For existing cohorts, patients should come from NUT-TB or NUSTART Cohorts
* For New HIV cohort, patients should be HIV positive ART naive, HIV negative participants will be come from the same neighborhood as newly recruited HIV positive patients
* Age will be 18 years and above
* Mwanza region residency
* Not planning to relocate outside Mwanza within the study period

Exclusion Criteria:

* Very severe illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective cohort study with two annual follow-ups will be conducted. This will be based on two existing HIV cohorts i.e. Nutrition, Diabetes and Pulmonary Tuberculosis (TB)/HIV (NUT-TB) (NCT00311298) conducted in Mwanza from 2006-2009 and Nutritional Support for African Adults Starting Antiretroviral Therapy (NUSTART) ( PACTR201106000300631) conducted in Mwanza during 2011-2013 and a new HIV cohort which will be recruited at study initiation. In the New HIV cohort, investigators will recruit both HIV patients and HIV negative participants who will act as controls. These 3 groups will provide about 1900 participants with and without HIV infection to address study objectives.
Sampling Method: Non-Probability Sample
Enrollment: 1947 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Combined prevalence of pre-diabetes and diabetes | Baseline and follow-up (12 and 24 months)
  The investigators will determine the combined prevalence of pre-diabetes and diabetes according to World Health Organization (WHO) diagnosis guidelines and investigate if behavioural and socio-demographic factors, and HIV, Tuberculosis (TB), ART, dyslipidaemia,chronic immune activation, parasitic infections, and body composition changes increase the risk of the outcome measure
Prevalence of hypertension | Baseline and follow-up (12 and 24 months)
  The investigators will determine the prevalence of hypertension according to WHO diagnosis guidelines and investigate if behavioural and socio-demographic factors, and HIV, TB, ART, dyslipidaemia,chronic immune activation, parasitic infections, and body composition changes increase the risk of the outcome measure

SECONDARY OUTCOMES:
Combined incidence of pre-diabetes and diabetes | Follow-up (12 and 24 months)
  The investigators will determine the combined incidence of pre-diabetes and diabetes. The number of patients meeting WHO diagnostic criteria of pre-diabetes and those meeting WHO diagnostic criteria for diabetes will added together and become the numerator whereas participants who are not pre-diabetic or diabetic at the beginning of the observation period will constitute the denominator. Investigators will determine if behavioural and socio-demographic factors, and HIV, TB, ART, dyslipidaemia,chronic immune activation, parasitic infections, and body composition changes increase the risk of the outcome measure
Prevalence of dyslipidaemia | Baseline and follow-up (12 and 24 months)
  The investigators will determine prevalence of dyslipidaemia based on WHO diagnosis guidelines and investigate if HIV and ART increase the risk of the outcome measure
Prevalence of diabetes clinical complications | Baseline and follow-up (12 and 24 months)
  The investigators will determine prevalence of diabetes clinical complications and investigate if HIV and ART increase or modify the risk of the outcome measure
Level of insulin resistance | Baseline and follow-up (12 and 24 months)
  The investigators will determine level of insulin resistance and investigate if HIV and ART are associated with the outcome measure
Level of beta-cell function | Baseline and follow-up (12 and 24 months)
  The investigators will determine level of beta-cell function and investigate if HIV and ART are associated with the outcome measure
Prevalence of diabetes by Fasting Blood Glucose (FBG), Oral Glucose Tolerance Test (OGTT) and Hba1c | Baseline
  By determining the prevalence of diabetes among HIV patients by 3 tests (FBG, OGTT and Hba1c), investigators will be able to judge the test which is best at diagnosing diabetes in HIV-infected populations.
Prevalence of sub-clinical atherosclerosis | Baseline and follow-up (12 and 24 months)
  The investigators will determine the prevalence of sub-clinical atherosclerosis and investigate if behavioural and socio-demographic factors, and HIV, TB, ART, dyslipidaemia,chronic immune activation, parasitic infections, and body composition changes increase the risk of the outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: George PrayGod, MD, PhD, Principal Investigator — National Institute for Medical Research (NIMR), Tanzania; Nyagosya Range, MSc, PhD, Principal Investigator — NIMR, Tanzania; Mette F Olsen, MSc, PhD, Principal Investigator — University of Copenhagen; Daniel Faurholt-Jepsen, MD, PhD, Principal Investigator — University of Copenhagen; Henrik Friis, MD, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- NIMR Research Clinic, Mwanza, Mwanza Region, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali MK, Magee MJ, Dave JA, Ofotokun I, Tungsiripat M, Jones TK, Levitt NS, Rimland D, Armstrong WS. HIV and metabolic, body, and bone disorders: what we know from low- and middle-income countries. J Acquir Immune Defic Syndr. 2014 Sep 1;67 Suppl 1:S27-39. doi: 10.1097/QAI.0000000000000256. PMID 25117959
- [Background] Tien PC, Schneider MF, Cole SR, Levine AM, Cohen M, DeHovitz J, Young M, Justman JE. Antiretroviral therapy exposure and incidence of diabetes mellitus in the Women's Interagency HIV Study. AIDS. 2007 Aug 20;21(13):1739-45. doi: 10.1097/QAD.0b013e32827038d0. PMID 17690572
- [Background] Florescu D, Kotler DP. Insulin resistance, glucose intolerance and diabetes mellitus in HIV-infected patients. Antivir Ther. 2007;12(2):149-62. doi: 10.1177/135965350701200214. PMID 17503657
- [Background] PrayGod G, Blevins M, Woodd S, Rehman AM, Jeremiah K, Friis H, Kelly P, Changalucha J, Heimburger DC, Filteau S, Koethe JR. A longitudinal study of systemic inflammation and recovery of lean body mass among malnourished HIV-infected adults starting antiretroviral therapy in Tanzania and Zambia. Eur J Clin Nutr. 2016 Apr;70(4):499-504. doi: 10.1038/ejcn.2015.221. Epub 2016 Jan 20. PMID 26785764
- [Background] Maganga E, Smart LR, Kalluvya S, Kataraihya JB, Saleh AM, Obeid L, Downs JA, Fitzgerald DW, Peck RN. Glucose Metabolism Disorders, HIV and Antiretroviral Therapy among Tanzanian Adults. PLoS One. 2015 Aug 19;10(8):e0134410. doi: 10.1371/journal.pone.0134410. eCollection 2015. PMID 26287742
- [Background] Dillon DG, Gurdasani D, Riha J, Ekoru K, Asiki G, Mayanja BN, Levitt NS, Crowther NJ, Nyirenda M, Njelekela M, Ramaiya K, Nyan O, Adewole OO, Anastos K, Azzoni L, Boom WH, Compostella C, Dave JA, Dawood H, Erikstrup C, Fourie CM, Friis H, Kruger A, Idoko JA, Longenecker CT, Mbondi S, Mukaya JE, Mutimura E, Ndhlovu CE, Praygod G, Pefura Yone EW, Pujades-Rodriguez M, Range N, Sani MU, Schutte AE, Sliwa K, Tien PC, Vorster EH, Walsh C, Zinyama R, Mashili F, Sobngwi E, Adebamowo C, Kamali A, Seeley J, Young EH, Smeeth L, Motala AA, Kaleebu P, Sandhu MS; African Partnership for Chronic Disease Research (APCDR). Association of HIV and ART with cardiometabolic traits in sub-Saharan Africa: a systematic review and meta-analysis. Int J Epidemiol. 2013 Dec;42(6):1754-71. doi: 10.1093/ije/dyt198. PMID 24415610
- [Background] PrayGod G, Changalucha J, Kapiga S, Peck R, Todd J, Filteau S. Dysglycemia associations with adipose tissue among HIV-infected patients after 2 years of antiretroviral therapy in Mwanza: a follow-up cross-sectional study. BMC Infect Dis. 2017 Jan 30;17(1):103. doi: 10.1186/s12879-017-2209-z. PMID 28137307
- [Derived] Nielsen ST, Kweka B, Praygod G, Filteau S, Olsen MF, Friis H, Faurholt-Jepsen D, Krogh-Madsen R. The incretin effect in type 2 diabetes in a Sub-Saharan African population. Clin Diabetes Endocrinol. 2024 Jul 25;10(1):20. doi: 10.1186/s40842-024-00178-5. PMID 39049087